CLINICAL TRIAL: NCT03820635
Title: Relation Between Plasma Concentration of Osteopontin Level and Vascular Calcification in Patients With Diabetic Nephropathy
Brief Title: Markers of Vascular Calcification in Diabetic Nephropathy in Patients With Diabetic Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud ahmed ali, Doctor, Assiut University
Other Study IDs: MVasCDN
Record Dates: First submitted 2019-01-26; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Diabetic Nephropathies; Vascular Calcification
MeSH Terms: conditions — Diabetic Nephropathies; Vascular Calcification

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Calcified: those with evidence of vascular calcification
  Interventions: Diagnostic Test: Osteopontin (OPN)
- Non-calcified: those with no evidence of vascular calcification
  Interventions: Diagnostic Test: Osteopontin (OPN)

INTERVENTIONS:
Diagnostic Test: Osteopontin (OPN) — the serum level of Osteopontin (OPN) will be measured in the subject's blood sample

SUMMARY:
The study will be conducted at Assiut University Hospital. Eligible subjects will be screened for vascular calcification by Doppler ultrasound examination. A correation between the level of serum Osteopontin (OPN) level and the extent of vascular calcification will be evaluated.

DETAILED DESCRIPTION:
Osteopontin (OPN) is one of integrin-binding N-linked glycoproteins, which is produced by activated mononuclear cells and is linked to increasing evidence about the role of OPN in vascular calcification[1].

Recent clinical studies have shown that vascular calcification is a pathological process leading to mechanical rigidity and stiffness of vascular wall, endothelial dysfunction, development and accelerating atherosclerosis even in the absence of established cardiovascular (CV) disease . Ectopic calcification is explained by several mutually counteracting molecular mechanisms, i.e. oxidative stress, microvascular inflammation, immune cell-to-cell cooperation, accumulation of lipids and extracellular proteins, vascular reparative systems, and metabolic disorders All these processes are under tight regulation of vitamin D, parathyroid hormone-related peptides (fibroblast growth factor, transcription factor Sox2, beta-catenin, etc) and matricellular proteins such as OPN. [2].

OPN was found to have relation with vascular calcification, atherosclerosis, and CV disease associated with severe vascular remodelling including hypertension, chronic kidney disease, diabetes mellitus . In this context, OPN is a promising biomarker of vascular remodelling closely related to inflammation intensity, glucose level and pro-thrombotic state with promising predictive value for CV events [3].

It is a matricellular protein that was first identified in 1995 by Heingard et al. as sialoprotein derived from bovine bone matrix . During the last decade a number of studies analysed the role of OPN in the pathogenesis of diabetic nephropathy. This proposed association needs confirmation and detailed description by further research [4].

At first, OPN has been reported to be highly expressed in the tubular epithelium of the renal cortex and in glomeruli in rat and mouse models of diabetic nephropathy [5]. This was associated with extensive macrophage accumulation in the kidney interstitium indicating that OPN upregulation and macrophage recruitment may play a role in the tubulo-interstitial injury in diabetic nephropathy [6]. Consistently, OPN/mice are protected from diabetes-induced albuminuria and renal damage, possibly by modulating podocyte signaling and motility [7]. In humans, plasma OPN levels are independently associated with presence and severity of diabetic nephropathy [8] Compelling evidence in the literature provides interesting clues about a link between the rennin-angiotensin system (RAS) and OPN in diabetic kidney disease. Diabetes-induced OPN expression and macrophage accumulation in the kidney interstitium of diabetic rats are significantly ameliorated after treatment with the long acting ACE inhibitor [9]. Showing that treatment with ramipril for nine month improves creatinine clearance rate and decreases urinary protein excretion, systolic blood pressure, development of glomerulosclerosis, tubulo-interstitial fibrosis and inflammatory cell infiltration in a diabetics. Of note, all these effects of ACE inhibition were associated with markedly suppressed OPN expression, suggesting that blockade of the RAS by ramipril may confer renoprotection by decreasing OPN secretion in diabetic nephropathy [10]. Liver X receptors (LXRs) have been identified as important lipid-dependent regulators of glucose metabolism and immune functions in leukocytes [11]. Synthetic LXR ligands can inhibit cytokine-induced OPN expression in macrophages [12]. Tachibana and colleges recently observed decreased urinary albumin excretion and substantially attenuated macrophage infiltration, mesangial matrix accumulation and interstitial fibrosis in streptozotocin-induced diabetics following administration of the LXR agonist T0901317. Notably, this was paralleled by diminished OPN expression in the kidney cortex indicating that inhibition of renal OPN by LXR activation may provide a potential therapeutical approach for diabetic nephropathy [13].

Osteopontin (OPN) is a multifunctional protein expressed by several different cell types, although the bone is known to be a major source [14].The exact excretion pathway of OPN from the body is not known. OPN is involved in a number of physiological and pathological conditions, including (1), urinary stones (2), wound healing (3), chronic inflammatory and autoimmune diseases (4), obesity-related chronic inflammation, and insulin resistance. However, OPN was originally found in bone and shown to regulate the formation and calcification of bone tissue. [15].

Notably, OPN has also been linked to vascular remodelling and calcification, especially in diabetic arteries, and has been shown to associate with diabetic retinopathy and nephropathy in patients with type 2 diabetes (T2D), as well as cardiovascular disease (CVD) events in diabetic subjects with history of long standing diabetes. [16]

ELIGIBILITY:
Inclusion Criteria:

* adult patients diagnosed clinically as diabetic nephropathy within 5 years

Exclusion Criteria:

* patients with any previous macrovascular complication: coronary heart disease, cerebrovascular stroke, peripheral ischaemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients diagnosed with diabetic nephropathies
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
correlation coefficient between serum level of osteoponton and the rate of different aspects of vascular affection as discussed previously | 6 months
  the correlation coefficient

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No